CLINICAL TRIAL: NCT00911833
Title: The Roles of Trust and Respect in Patient Reactions to Race-Based and Personalized Medicine Vignettes: An Experimental Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909153; 09-HG-N153
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-30

CONDITIONS: Diabetes; Congenital Heart Disease; Hypertension
Keywords: Trust
MeSH Terms: conditions — Diabetes Mellitus; Heart Defects, Congenital; Hypertension

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Genetic research has implications for drug development and marketing. Race-based medicine may be able to provide specific treatment for populations with increased disease-specific morbidity and mortality. However, contemporary genetic research refutes the idea that races are genetically distinct populations, even as drugs designed for use in specific races are being promoted.
* Studies have shown high levels of public suspicion for race-based and personalized genetic medicine. Concerns related to not only the potential performance of race-based drugs, but also the motives of those offering these drugs. Many participants have suggested conspiracy theories in which race-based medicine was disguising an attempt to provide inferior medications or deliberately harm certain populations. Concerns about personalized medicine often have to do with privacy and other personal concerns.
* Public suspicions of race-based medicine, and to a lesser extent, personalized genetic medicine, make it important to examine and understand the theoretical and empirical literature on trust and health care.

Objective:

- To describe the perspective of participants evaluating the medicine offer.

Eligibility:

* Males and females ages 18 and older who are visiting the John Hopkins clinics (primarily the adult care clinics).
* Participants must be able to take a literacy screen and respond to a short survey.

Design:

* Participants will be asked to take a researcher-administrated literacy screen, read one of three randomly assigned vignettes, and fill out a survey. The first page of the survey will provide information about the study.
* Participants will respond to initial questions about demographics, experiences with discrimination, and trust in the medical profession and institutions.
* Each participant will receive a random vignette in which he/she will imagine him/herself being diagnosed with a common, chronic condition and offered a conventional drug, a race-based drug, or a genetically personalized drug.
* After being presented with the vignette, participants will be asked to respond to a survey that asks about their levels of trust in the vignette doctor, perceived respect given to the patient by the vignette physician, emotional response to the vignette, their belief in the effectiveness and safety of the drug prescribed in the vignette, information sufficiency, and their hypothetical behavioral intention to take the drug.
* Participants will be debriefed after completing the survey, and will be offered a small amount of compensation for participating.

DETAILED DESCRIPTION:
This study proposes to describe participants' attitudinal, emotional, cognitive, and hypothetical behavioral responses to randomized hypothetical vignettes illustrating the prescription of conventional, race-based, and genetically personalized medicine for a common chronic condition. This study is theoretically guided by conceptualizations of relationship-centered care and the risk information seeking and processing model. These theories recognize the importance of interpersonal influence within health care interactions, underscore the moral dimensions of patient-physician relationships, and describe the predictors of how information is attended to and processed. An experimental, mixed methods design will be used to randomly assign 357 patients at the Johns Hopkins clinics to one of three vignettes illustrating conventional, race-based, and genetically personalized medication offers. This study aims to examine the effects of the type of medication offer (conventional, race-based, and genetically personalized) and certain participant characteristics (race, literacy, background healthcare trust/experience with discrimination) on attitudinal, emotional, cognitive, and hypothetical behavioral responses; to determine if the relationships among the type of medication offer and the four categories of outcomes are moderated by race and mediated by trust; and to describe the participants' perspective on the vignette, through targeted open-ended questions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants are primarily African American or white, have a high prevalence of chronic disease, and a moderate prevalence of limited literacy.

Participants must be 18 or older.

EXCLUSION CRITERIA:

Participants who do not speak English and cannot read the survey (due to linguistic barriers) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-05-19; Study Completion 2011-03-30

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beach MC, Roter DL, Wang NY, Duggan PS, Cooper LA. Are physicians' attitudes of respect accurately perceived by patients and associated with more positive communication behaviors? Patient Educ Couns. 2006 Sep;62(3):347-54. doi: 10.1016/j.pec.2006.06.004. Epub 2006 Jul 21. PMID 16859867
- [Background] Beach MC, Sugarman J, Johnson RL, Arbelaez JJ, Duggan PS, Cooper LA. Do patients treated with dignity report higher satisfaction, adherence, and receipt of preventive care? Ann Fam Med. 2005 Jul-Aug;3(4):331-8. doi: 10.1370/afm.328. PMID 16046566
- [Background] Bevan JL, Lynch JA, Dubriwny TN, Harris TM, Achter PJ, Reeder AL, Condit CM. Informed lay preferences for delivery of racially varied pharmacogenomics. Genet Med. 2003 Sep-Oct;5(5):393-9. doi: 10.1097/01.gim.0000087989.12317.3f. PMID 14501835